CLINICAL TRIAL: NCT05488327
Title: Safety and Efficacy of Lenalidomide in the Treatment of Refractory Cutaneous Dermatomyositis
Brief Title: Lenalidomide in the Treatment of Refractory Cutaneous Dermatomyositis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangxi Provincial People's Hopital (Other)
Responsible Party: Principal Investigator, Lihua Duan, Dr, Jiangxi Provincial People's Hopital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLH88086
Record Dates: First submitted 2022-07-28; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Dermatomyositis
Keywords: Cutaneous Dermatomyositis, Lenalidomide
MeSH Terms: conditions — Dermatomyositis | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention with lenalidomide (Experimental): All subjects will be treated with lenalidomide 5mg/day.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — All subjects will be treated with lenalidomide 5mg/day with a regular follow-up of 24 weeks.

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of lenalidomide in the treatment of patients with active cutaneous DM.

DETAILED DESCRIPTION:
Dermatomyositis (DM) are systemic immune-mediated inflammatory diseases which commonly affected the skin and musculoskeletal system. The cutaneous manifestations of DM are the most important aspect of this disease. Treatment of these cutaneous manifestations is challenging and currently no universally effective drugs exists. Lenalidomide, a second-generation derivative of thalidomide, has a role as an angiogenesis inhibitor, an antineoplastic agent and an immunomodulator. Reports on refractory cutaneous manifestations of systemic lupus erythematosus have been mostly performed. The clinical trials of lenalidomide for cutaneous DM are lacking. This is a single-centre, prospective, open-label, single-arm study with Lenalidomide 5mg/day added to the background treatment of GCs and immunosuppressants in DM to evaluate the efficacy and safety of lenalidomide in the treatment of cutaneous DM.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant、non-nursing female.
2. Age 18 to 75 years at the time of signing informed consent.
3. Fulfilling 2017 ACR/EULAR IIMs classification criteria for DM or ADM.
4. Disease activity with skin damage (CDASI ≥12) despite treatment with corticosteroids, immunosuppressive agents or biologics for more than 3 months.
5. Written informed consent obtained before taking part in the study.

Exclusion Criteria:

1. Pregnant women or breastfeeding mothers, Male and female patients with recent fertility requirements.
2. Skin and mucosal lesions should exclude erythema multiforme, syphilis, Sweet disease, Stevens-Johnson syndrome, acne vulgaris, herpes simplex infection, periodic granulocytopenia, and acquired immunodeficiency.
3. Severe Concomitant disease: including heart failure (≥level Ⅲ, NYHA), respiratory failure, myelosuppression (WBC<3.0×109/L or N<1.5×109/L, HGB≤85g/L, PLT<100×109/L), peripheral neuropathy.
4. Acute severe infections such as sepsis and cellulitis, active hepatitis B or C virus infection, active tuberculosis, and history of a positive test for, or any clinical suspicion of, human immunodeficiency virus (HIV).
5. Patients with risk factors for myocardial infarction (including a history of thrombosis), hypercoagulability, or with history of venous thromboembolism, including deep vein thrombosis and pulmonary embolism.
6. Patients with allergies or contraindications to lenalidomide or thalidomide.
7. Uncontrolled or rapidly progressive myositis or interstitial lung disease at the discretion of the investigator which is likely to warrant escalation in therapy beyond permitted background medications.
8. Recurrent or chronic bacterial, viral, fungal, mycobacterial, or other infections including HIV.
9. History of recurrent herpes zoster, disseminated (multi-dermatomal) herpes zoster, disseminated herpes simplex or ophthalmic zoster. Herpes zoster lesions within 90 days prior to screening.
10. Primary or secondary immunodeficiency.
11. Current uncontrolled renal, gastrointestinal, endocrine, pulmonary, cardiac, or neurologic disease, which, in the opinion of the investigator, might place the patient at unacceptable risk for participation in this study.
12. History of alcohol, drug, or chemical abuse within one year prior to signing the informed consent form.
13. Major surgery within 8 weeks prior to Screening or planned major surgery at any time during participation in the study.
14. Immunization with a live/attenuated vaccine within 4 weeks prior to Screening.
15. History of malignant tumor within 5 years prior to screening (stable disease for more than 6 months after completion of tumor treatment program can be enrolled).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Cutaneous Disease Activity Severity Index (CDASI) activity score | 24 weeks
  Change in Cutaneous Disease Activity Severity Index (CDASI) activity score (0-100), higher scores mean a worse outcome

SECONDARY OUTCOMES:
Cutaneous Disease Activity Severity Index (CDASI) activity score | 12 weeks
  Change in Cutaneous Disease Activity Severity Index (CDASI) activity score (0-100), higher scores mean a worse outcome
International Myositis Assessment & Clinical Studies Group (IMACS) Disease Activity Core Set Measures | 12 weeks and 24 weeks
  Change in International Myositis Assessment & Clinical Studies Group (IMACS) Disease Activity Core Set Measures
SF-36 | 12 weeks and 24 weeks
  Change in SF-36
Dermatology Life Quality Index (DLQI) | 12 weeks and 24 weeks
  Change in Dermatology Life Quality Index (DLQI)
Adverse event | 24 weeks
  Adverse event monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Lihua Duan, MD, Principal Investigator — Jiangxi Provincial People's Hopital
Locations (1):
- Department of Rheumatology and Clinical Immunology, Jiangxi Provincial People's Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No